CLINICAL TRIAL: NCT00087581
Title: An Open-Label, Prospective, Randomized, Controlled, Multi-Center Study Assessing Fixed Dose Versus Concentration Controlled Cellcept® Regimens for Patients Following a Single Organ Renal Transplantation in Combination With Full Dose and Reduced Dose Calcineurin Inhibitors
Brief Title: Study of Therapeutic Monitoring of Mycophenolate Mofetil (MMF/CellCept) After Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML17225
Record Dates: First submitted 2004-07-12; First posted 2004-07-14 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Mycophenolic Acid; Cyclosporine; Tacrolimus

ARMS (3):
- Group A: Monitored MMF + Reduced CNI (Experimental): Group A will receive concentration-controlled/monitored MMF with an oral CNI, either cyclosporine or tacrolimus. Depending on body surface area and age, MMF may be given in capsule, tablet, oral suspension, or intravenous (IV) form. The initial dose will be at least 1 gram twice a day (BID) in adults and 600 milligrams per meter-squared (mg/m^2) in pediatrics. Subsequent doses will be adjusted to maintain blood mycophenolic acid (MPA) levels greater than or equal to (≥) 1.3 micrograms per milliliter (μg/mL) with cyclosporine or ≥1.9 μg/mL with tacrolimus. The selected CNI will be dosed to maintain reduced blood concentrations. Cyclosporine target concentrations are as follows: Days 1-30, 250-325 nanograms per milliliter (ng/mL); Days 30-90, 125-165 ng/mL; Days 90 through end of study, 95-145 ng/mL. Tacrolimus target concentrations areas follows: Days 1-30, 8-12 ng/mL; Days 30-90, 4-6 ng/mL; Days 90 through end of study, 3-5 ng/mL.
  Interventions: Drug: Mycophenolate mofetil; Drug: Cyclosporine; Drug: Tacrolimus
- Group B: Monitored MMF + Full CNI (Experimental): Group B will receive concentration-controlled/monitored MMF with an oral CNI, either cyclosporine or tacrolimus. Depending on body surface area and age, MMF may be given in capsule, tablet, oral suspension, or IV form. The initial dose will be at least 1 gram BID in adults and 600 mg/m^2 in pediatrics. Subsequent doses will be adjusted to maintain blood MPA levels ≥1.3 μg/mL with cyclosporine or ≥1.9 μg/mL with tacrolimus. The selected CNI will be dosed to maintain standard/full blood concentrations. Cyclosporine target concentrations are as follows: Days 1-30, 250-325 ng/mL; Days 30-90, 250-270 ng/mL; Days 90 through end of study, 190-220 ng/mL. Tacrolimus target concentrations are as follows: Days 1-30, 8-12 ng/mL; Days 30-90, 8-10 ng/mL; Days 90 through end of study, 6-8 ng/mL.
  Interventions: Drug: Mycophenolate mofetil; Drug: Cyclosporine; Drug: Tacrolimus
- Group C: Fixed MMF + Full CNI (Experimental): Group C will receive fixed-dose MMF with an oral CNI, either cyclosporine or tacrolimus. Depending on body surface area and age, MMF may be given in capsule, tablet, oral suspension, or IV form. The dose will be at least 1 gram BID in adults and 600 mg/m^2 in pediatrics. Subsequent doses are not to be adjusted, except in the case of unacceptable toxicity. The selected CNI will be dosed to maintain standard/full blood concentrations. Cyclosporine target concentrations are as follows: Days 1-30, 250-325 ng/mL; Days 30-90, 250-270 ng/mL; Days 90 through end of study, 190-220 ng/mL. Tacrolimus target concentrations are as follows: Days 1-30, 8-12 ng/mL; Days 30-90, 8-10 ng/mL; Days 90 through end of study, 6-8 ng/mL.
  Interventions: Drug: Mycophenolate mofetil; Drug: Cyclosporine; Drug: Tacrolimus

INTERVENTIONS:
Drug: Mycophenolate mofetil — Depending on body surface area and age, MMF may be given in capsule, tablet, oral suspension, or IV form. The initial dose will be at least 1 gram BID in adults and 600 mg/m^2 in pediatrics. In Groups A and B, subsequent doses will be adjusted to maintain blood MPA levels ≥1.3 μg/mL with cyclosporine or ≥1.9 μg/mL with tacrolimus. In Group C, subsequent doses are not to be adjusted, except in the case of unacceptable toxicity.
  Other Names: CellCept
Drug: Cyclosporine — Cyclosporine will be given as 100-mg soft gelatin capsules and dosed to maintain either reduced (Group A) or standard/full (Groups B and C) blood concentrations. Cyclosporine target concentrations are as follows: Days 1-30, 250-325 ng/mL; Days 30-90, 125-165 ng/mL (reduced) or 250-270 ng/mL (full); Days 90 through end of study, 95-145 ng/mL (reduced) or 190-220 ng/mL (full).
  Other Names: Neoral
Drug: Tacrolimus — Tacrolimus will be given as 1-mg and 5-mg capsules and dosed to maintain either reduced (Group A) or standard/full (Groups B and C) blood concentrations. Tacrolimus target concentrations are as follows: Days 1-30, 8-12 ng/mL; Days 30-90, 4-6 ng/mL (reduced), 8-10 ng/mL (full); Days 90 through end of study, 3-5 ng/mL (reduced), 6-8 ng/mL (full).
  Other Names: Prograf

SUMMARY:
This three-arm study will evaluate the efficacy and safety of various dosing regimens of MMF combined with various dosing regimens of calcineurin inhibitor (CNI), either cyclosporine or tacrolimus, in participants who have undergone kidney transplantation. Participants will be randomized to one of three dosing regimens to receive concentration-controlled MMF with reduced CNI, concentration-controlled MMF with standard CNI, or fixed-dose MMF with standard CNI. Participants will be followed for 20-24 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 13-75 years of age
* Single organ recipient (kidney only) from living (related or unrelated) or cadaveric heart-beating donors
* Receiving first or second kidney transplant

Exclusion Criteria:

* Immunosuppressive therapy (except for 48 hours prior to transplantation and corticosteroid treatment) within previous 28 days for a first transplant and 3 months for a second transplant
* History of malignancy in last 5 years (except successfully treated localized non-melanoma skin cancer)

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2004-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Treatment Failure During 12 Months Post-Transplantation | Month 12
Percent Change from Baseline in Calculated Glomerular Filtration Rate (GFR) at 12 Months Post-Transplantation | Baseline to Month 12

SECONDARY OUTCOMES:
Percentage of Participants with Treatment Failure During 6 and 20-24 Months Post-Transplantation | Months 6, 20-24
Percentage of Participants with Biopsy-Proven Acute Rejection (BPAR) | Months 6, 12, 20-24
Percentage of Participants by Number of BPAR Episodes | Months 6, 12, 20-24
Percentage of Participants Treated for Acute Rejection (AR) | Months 6, 12, 20-24
Percentage of Participants Who Experienced Graft Loss | Months 6, 12, 20-24
Percentage of Participants Who Died | Months 6, 12, 20-24
Percentage of Participants Who Discontinued Treatment with MMF | Months 6, 12, 20-24
Time to First BPAR Episode | Months 6, 12, 20-24
Time to Treatment Failure | Months 6, 12, 20-24
Percent Change from Baseline in Calculated GFR at 3, 6, and 20-24 Months Post-Transplantation | Baseline to Months 3, 6, 20-24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (51):
- United States (51):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Bakersfield, California
  - Los Angeles, California
  - San Francisco, California
  - Denver, Colorado
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Springfield, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Rochester, Minnesota
  - Hackensack, New Jersey
  - Livingston, New Jersey
  - Buffalo, New York
  - Hawthorne, New York
  - New York, New York
  - Rochester, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cleveland, Ohio
  - Portland, Oregon
  - Harrisburg, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Falls Church, Virginia
  - Norfolk, Virginia
  - Seattle, Washington
  - Madison, Wisconsin